CLINICAL TRIAL: NCT06287645
Title: Development of Digital Fundus Images Dataset of Local Population of Pakistan
Brief Title: Color Fundus Photograph With Experts Labelling
Status: Recruiting | Type: Observational
Sponsor: Pakistan Council of Scientific and Industrial Research (Other)
Collaborators: Al-Ibrahim Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Retinal Images Dataset
Record Dates: First submitted 2024-02-21; First posted 2024-03-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Retinal Disease; Diabetic Retinopathy
MeSH Terms: conditions — Retinal Diseases; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Color Fundus Photography/Non-Mydriatic Opthalmic Cameras — Participants will undergo retinal imaging by fundus camera. Three specialists will independently grade images for common retinal disorders like Diabetic Retinopathy. Final grading decisions will be unanimous among the specialists.

SUMMARY:
This trial aims to provide a digital retinal image dataset from Pakistan, graded by three specialists according to the severity of Diabetic Retinopathy. The dataset aims to improve research and patient care.

DETAILED DESCRIPTION:
This clinical trial aims to address the scarcity of retinal image datasets in Pakistan by providing a comprehensive digital fundus photograph dataset, accompanied by expert grading. The dataset will encompass retinal images from Pakistani individuals, meticulously labeled by three Vitreo Retinal Specialists. These specialists will assess the presence and severity of common retinal disorders, including No Diabetic Retinopathy (No DR), Mild, Moderate, Severe, Proliferative Diabetic Retinopathy, Clinically Significant Macular Edema (CSME), and Advance diabetic Eye Diseases (ADED). Each image will also be evaluated for diagnostic clarity and the presence of any additional findings. Final grading decisions will be reached through unanimous consensus among the graders, ensuring the dataset's reliability and accuracy. This initiative holds promise for advancing ophthalmic research and improving patient care in Pakistan and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type I or Type II Diabetes.
* Patients of age of 20 years or above

Exclusion Criteria:

* The participant is unable or unwilling to comply with study procedures.
* Vulnerable participants (minors, legally detained individuals).
* Prisoners or subjects who are involuntarily incarcerated.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the diabetic eye care center at our collaborated hospital will be registered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Grading Diabetic Retinopathy Severity according to International Clinical Diabetic Retinopathy Severity Scale | 1 Visit (1 day)
  Each Fundus photograph will be evaluated according to the Severity of Diabetic Retinopathy following International Clinical Diabetic Retinopathy Severity Scale (ICDRSS). Following Diabetic Retinopathy symptoms will be graded according to this scale.
  1. No DR
  2. Mild
  3. Moderate
  4. Severe
  5. Proliferative
Grading Diabetic Retinopathy Severity according to Early Treatment of Diabetic Retinopathy Scale | 1 Visit (1 day)
  Each Fundus photograph will be evaluated according to the Severity of Diabetic Retinopathy following Early Treatment of Diabetic Retinopathy Scale (ETDRS). Following Diabetic Retinopathy symptoms will be graded according to this scale.
  1. Clinically Significant Macular Edema
  2. Advance Diabetic Eye Disease
Finding inter-rater agreement among the graders | Two Years
  The intraclass correlation coefficient will be calculated using the collected dataset to assess the consistency in grading among all graders.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Mustafa, Principal Investigator — Pakistan Council of Scientific and Industrial Research
Locations (1):
- Al Ibrahim Eye Hospital, Karachi, Pakistan